CLINICAL TRIAL: NCT07033624
Title: Cardiovascular Risk Early Screening and Warning in Harbin : A Prospective Cohort Study
Status: Not yet recruiting | Type: Observational
Sponsor: Harbin Medical University (Other)
Responsible Party: Principal Investigator, Yu Bo, Director, Cardiology Department, the 2nd Affiliated Hospital of Harbin Medical University, Harbin Medical University
Other Study IDs: KY2025-042
Record Dates: First submitted 2025-06-13; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Cardiovascular Diseases
Keywords: Cardiovascular diseases, microbiome, genomics, metabolism, imaging, risk prediction
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this prospective cohort study is to collect the multi-omics profile of cardiovascular disease (CVD) high-risk individuals in Harbin, and to discover novel biomarker signatures of major adverse cardiovascular events (MACE) during a minimum 2-year follow-up period.

DETAILED DESCRIPTION:
This is a single-center, observational, prospective cohort study. The primary endpoint is the incidence of MACE. Participants must meet at least two of the following criteria: hypertension, hyperglycemia, hyperlipidemia, or obesity. Baseline data and biological samples will be collected at enrollment, with clinical outcomes monitored for a minimum of two years. The study aims to enroll 10,000 participants aged 45 years and older from Harbin city, located in northeastern China.

ELIGIBILITY:
Inclusion Criteria:

* 1.Residents of Harbin city, regardless of gender.
* 2.Meets at least two of the following conditions: diabetes, hypertension, hyperlipidemia, or obesity.
* 3.No history of cardiovascular or cerebrovascular diseases.
* 4.Willing to participate in the study and sign the informed consent form

Exclusion Criteria:

* 1.History of antibiotic or probiotic treatment within the past month.
* 2. Pregnant women.
* 3. History of autoimmune diseases or malignant tumors; severe heart, liver, or kidney dysfunction; or a history of severe cardiovascular or cerebrovascular diseases.
* 4. Any unstable condition or situation that may jeopardize patient safety or compliance.
* 5. Patients unable to provide informed consent due to physical reasons or unwilling to participate.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will enroll 10,000 participants aged 45 and above from Harbin, a city in northeastern China. To be eligible, participants must meet at least two of the following criteria: hypertension, hyperglycemia, hyperlipidemia, or obesity.
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2047-07-01 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiovascular event (MACE) | 2 years
  A major adverse cardiovascular event (MACE) of cardiovascular death, nonfatal myocardial infarction, and nonfatal stroke

SECONDARY OUTCOMES:
Cardiovascular death | 2 years
  Cardiovascular death
All-cause death | 2 years
  All-cause death
Myocardial infarction | 2 years
  Myocardial infarction
Stroke | 2 years
  Stroke

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang, China